CLINICAL TRIAL: NCT05980468
Title: The Effect of Music Therapy on Nurses' Comfort Levels
Brief Title: The Effect of Music Therapy on Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Assistant Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 05/2023
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Music Therapy
Keywords: nurse; comfort; music therapy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Music intervention sessions will be applied to each participant for 5 weeks, 3 days a week, 20 minutes per session. Forms will be applied at the first meeting and for five weeks.
  Interventions: Other: music therapy
- Control group (No Intervention): No application has been made. Forms will be applied at the first meeting and for five weeks.

INTERVENTIONS:
Other: music therapy — Music intervention sessions will be applied to each participant for 5 weeks, 3 days a week, 20 minutes per session.
  Arms: Intervention group

SUMMARY:
This study was planned to examine the effect of music therapy on the comfort levels of nurses. In the study, data will be collected by using Descriptive Characteristics Information Form and Nurse Comfort Scale. Whether the nurses who meet the inclusion criteria will be in the intervention or control group will be determined by simple randomization. Music intervention sessions will be applied to each participant for 5 weeks, 3 days a week, 20 minutes per session. After 5 weeks, the Nurse Comfort Scale will be applied to the participants again.

DETAILED DESCRIPTION:
This study was planned to examine the effect of music therapy on the comfort levels of nurses. This study will be conducted as a randomized controlled experimental study. In the sample calculation, it was determined that for Power = 0.8 (beta = 0.2), alpha = 0.05 and effect size = 0.7, the sample size should be 66, 33 for the intervention group and 33 for the control group. In the study, data will be collected by using Descriptive Characteristics Information Form and Nurse Comfort Scale. Whether the nurses who meet the inclusion criteria will be in the intervention or control group will be determined by simple randomization. Music intervention sessions will be applied to each participant for 5 weeks, 3 days a week, 20 minutes per session. After 5 weeks, the Nurse Comfort Scale will be applied to the participants again. Research data will be analyzed in SPSS-25 package program.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one year of working experience
* Have not participated in any music therapy session before
* No hearing problems
* Absence of neurological/psychiatric disorders
* Nurses who volunteered to participate in the study will be included in the study.

Exclusion Criteria:

* Those who use another relaxation methods,
* Nurses who do not agree to participate in the study will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Comfort | 5 weeks after first meeting
  The scale consists of 39 items in total. Each statement in the scale has a Likert-type rating ranging from 1-4 from "strongly disagree" to "strongly agree". 24 of the expressions are positive and 15 are negative, and negative items are reversed in scoring. Accordingly, a high score (4) indicates high comfort, a low score (1) indicates low comfort, and a low score (1) indicates high comfort in negative statements, and a high score (4) indicates low comfort. The Cronbach alpha coefficient was found to be 0.915.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Korkut, Principal Investigator — TC Erciyes University; Ayşe Topuz, Principal Investigator — Karamanoğlu Mehmetbey University
Locations (1):
- Sevda Korkut, Talas, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No